

Version Date: Version 3 (3/16/2022)

| Destining and Manage | Data |
|---|---|
| Participant Name: | Date: |
| Title of Study: Highly challenging balance program to reduce fall rate in PD | |
| Principal Investigator: Dr. David Sparrow | VA Facility: VA Boston Healthcare System |

#### **KEY SUMMARY INFORMATION ABOUT THIS STUDY**

We are asking you to be in a research study that is being supported by the VA Office of Rehabilitation Research and Development. Before you decide to take part, you should know why the study is being done and what it will involve. This form tells you what to expect if you agree to be in the study. Taking part in this study is completely voluntary; it is your decision whether or not to participate in the study.

## WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

We are doing the research to evaluate the effect of exercise on balance and fall rate. If you agree, you will complete some questionnaires and a balance assessment and participate in one of three programs. You will be in the study for 6 months if you decide to stay for the whole study. We will describe your involvement in more detail later in this form.

## WHAT ARE KEY REASONS YOU MIGHT CHOOSE TO VOLUNTEER FOR THIS STUDY?

You might choose to volunteer in the study because the program might potentially improve your balance, physical fitness, and quality of life. For a complete description of benefits, refer to the Detailed Information section of this form.

# WHAT ARE KEY REASONS YOU MIGHT CHOOSE NOT TO VOLUNTEER FOR THIS STUDY?

You may choose not to volunteer to be in the study because of the possibility that you may experience discomfort during normal exercise. For a complete description of risks, refer to the Detailed Information section of this form.

#### DO YOU HAVE TO TAKE PART IN THE STUDY?

If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits or rights you would normally have if you choose not to volunteer.

## WHAT IF YOU HAVE QUESTIONS, SUGGESTIONS OR CONCERNS?

The person in charge of the study is Dr. David Sparrow at the VA Boston Healthcare System. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study, his contact information is 857-364-6400

FOR IRB USE ONLY

VA Boston Healthcare System IRB
Effective Date: April 11, 2022



Version Date: Version 3 (3/16/2022)

| Participant Name: | Date: |
|---|---|
| Title of Study: Highly challenging balance program to reduce fall rate in PD | |
| Principal Investigator: <b>Dr. David Sparrow</b> | VA Facility: VA Boston Healthcare System |

#### **DETAILED INFORMATION ABOUT THE STUDY**

## WHAT IS THE PURPOSE OF THIS STUDY?

The purpose of this research study is to compare different approaches to providing a safe exercise program to people with Parkinson's disease.

#### **HOW LONG WILL I BE IN THE STUDY?**

We are asking you and approximately 162 veterans to participate in this study. This research study is expected to take approximately 4 years to complete. Your individual participation in the project will take 6 months.

## WHAT WILL HAPPEN IF I TAKE PART IN THE STUDY?

You will be allowed to participate as long as your physician has no objections to your participation. You will be asked to complete three evaluations over a 6-month period (at baseline, 3 months, and 6 months) at the Jamaica Plain campus of the VA Boston Healthcare System. We may ask you to complete the consent process over the phone before you come in for your visit.

At the first evaluation (baseline), you will be asked to complete some questionnaires and undergo some balance assessments. The questionnaires will take approximately 20 minutes and will be completed over the phone during a scheduled call or in person at the Jamaica Plain campus of the VA Boston Healthcare System. The balance assessments will take place at the Jamaica Plain campus of the VA Boston Healthcare System and will take approximately 30 minutes. If you meet all eligibility criteria, you subsequently will be randomly assigned – that is, by chance – to one of three groups. You will be shipped at no cost to you all study materials and equipment based on your assigned group.

If assigned to the first group, you will be asked to carry out a structured weekly exercise program at the Jamaica Plain campus of the VA Boston Healthcare System for 3 months. The exercise sessions will be scheduled two times per week for 1.5 hours each session; however, during periods that face-to-face time with study staff needs to be reduced, sessions will be scheduled three times per week for 1 hour each session.

If assigned to the second group, you will be asked to carry out a structured exercise program in your home following instructions on a smartphone 3 times per week for 3 months. Also, during some of your sessions, we will observe you remotely while you exercise using VA Video Connect. A typical session will last about one hour.

FOR IRB USE ONLY



Version Date: Version 3 (3/16/2022)

| Participant Name: | |
|---|---|
| Title of Study: Highly challenging balance program to reduce fall rate in PD | |
| Principal Investigator: Dr. David Sparrow | VA Facility: VA Boston Healthcare System |

If assigned to the third group, you will be taught a lifestyle exercise program in which you will hear about similar exercises and, in addition, will be advised about general health topics for 3 months. You will use a smartphone 3 times per week to listen to this information. A typical session will last about 15 minutes.

You will also be asked to complete a diary each week during the 6 months to record any falls you might have.

At 3 months and again at 6 months, you will be asked to repeat the balance assessments and repeat the questionnaires. The questionnaires will take approximately 20 minutes and may be completed over the phone or in person at the Jamaica Plain campus of the VA Boston Healthcare System. The balance assessments will take place at the Jamaica Plain campus of the VA Boston Healthcare System and will take approximately 30 minutes.

During your 6 months of participation, we will call you every 2 weeks to check on how you are doing. When your participation is complete, you will be asked to ship all study equipment back to us at no cost to you.

#### WHAT IS EXPECTED OF ME IF I TAKE PART IN THIS STUDY?

- Keep your study appointments. If you miss an appointment, please contact the investigator or research staff to reschedule as soon as you know you will miss the appointment.
- Complete your questionnaires as instructed.
- Ask questions as you think of them.
- Tell the investigator or research staff if you believe you might be pregnant or might have gotten your partner pregnant.
- While participating in this research study, do not take part in any other research project without
  approval from the investigators. This is to protect you from possible injury from things such as extra
  blood drawing, extra X-rays, or potential drug interactions. Taking part in other research studies
  without first discussing it with the investigators of this study may invalidate the results of this study, as
  well as that of the other studies.

## WHAT POSSIBLE RISKS OR DISCOMFORTS MIGHT I HAVE IF I TAKE PART IN THIS STUDY?

Any procedure has possible risks and discomforts. The procedures in this study may cause all, some, or none of the risks or side effects listed. Rare, unknown, or unexpected risks also may occur.

Discomfort or inconvenience involved in this study are those associated with normal mild exercise. You may experience fatigue as your muscles tire or ache during or immediately after exercising.

FOR IRB USE ONLY

VA Boston Healthcare System IRB

Effective Date: April 11, 2022



Version Date: Version 3 (3/16/2022)

| Participant Name: | Date: |
|---|---|
| Title of Study: Highly challenging balance program to reduce fall rate in PD | |
| Principal Investigator: <b>Dr. David Sparrow</b> | VA Facility: VA Boston Healthcare System |

The risks associated with training include strained and pulled muscles, rapid heart beat, labored breathing, chest discomfort, light-headedness, dizziness and falls. If you experience any of these symptoms, you should stop exercising and contact your physician as well as study staff.

Also, in addition to the risks listed above, you may experience a previously unknown risk or side effect.

If you are or become pregnant, the particular treatment or procedure might involve risks to the embryo or fetus, which are currently unforeseeable.

## WHAT ARE THE POSSIBLE BENEFITS OF THIS STUDY?

There are no direct/personal benefits to you from your taking part in this research study. However, the information we get from this study might help others with your condition.

#### **HOW WILL MY PRIVATE INFORMATION BE PROTECTED?**

Taking part in this study will involve collecting private information about you. This information will be protected in the following ways:

To protect confidentiality, data will be identified only by study ID number assigned to you. All computer files will be secured using access permissions and assigned passwords to ensure only authorized study personnel will have access to your data. Access permissions and passwords will be changed whenever there has been a change in study personnel. Any required personal information on you will be kept in a separate file and only the Principal Investigator and Study Coordinator will have access permissions granted to this file. All of your paper forms will be secured in a locked fireproof study cabinet. Only the Principal Investigator will have keys to the study cabinet.

There are times when we might have to show your records to other people. For example, someone from the Office of Human Research Protections, the Government Accountability Office, the Office of the Inspector General, the VA Office of Research Oversight, the VA Institutional Review Board (IRB), our local Research and Development Committee, and other study monitors may look at or copy portions of records that identify you.

Your information collected as part of the research, even if identifiers are removed, will not be used or distributed for future research studies.

FOR IRB USE ONLY



Version Date: Version 3 (3/16/2022)

| Participant Name: | Date: |
|---|---|
| Title of Study: Highly challenging balance program to reduce fall rate in PD | |
| Principal Investigator: Dr. David Sparrow | VA Facility: VA Boston Healthcare System |

## **Health Information Portability and Accountability Act (HIPAA)**

There are rules to protect your private information. Federal and state laws and the federal medical Privacy Rule also protect your privacy. By signing this form, you provide your permission called your 'authorization,' for the use and disclosure of information protected by the HIPAA Privacy Rule.

The research team working on the study will collect information about you. This includes things learned from the procedures described in this consent form. The study team may also collect other information including your name, address, date of birth, and information from your medical records such as your medical history.

The research team may also need to disclose the information to others as part of the study progress. Others may include the following: the Institutional Review Board, Research & Development Committee, Research Compliance Officers, Office of Human Research Protections (OHRP), the VA Office of Research Oversight (ORO), and the Government Accountability Office (GAO) and the local VA medical facility Human Research Protections Program.

Your health information disclosed pursuant to this authorization may no longer be protected by Federal laws or regulations and may be subject to re-disclosure by the recipient.

While this study is being conducted you will not have access to your research related health records.

This will not affect your VA healthcare, including your doctor's ability to see your records as part of your normal care and will not affect your right to have access to the research records after the study is completed.

You can revoke this authorization, in writing, at any time. To revoke your authorization, you must write to the Release of Information Office at this facility or you can ask a member of the research team to give you a form to revoke the authorization. Your request will be valid when the Release of Information Office receives it. If you revoke this authorization, you will not be able to continue to participate in the study. This will not affect your rights as a VHA patient to treatment or benefit outside of the study.

If you revoke this authorization, Dr. David Sparrow and his research team can continue to use information about you that was collected before receipt of the revocation. The research team will not collect information about you after you revoke the authorization.

Treatment, payment or enrollment/eligibility for benefits cannot be conditioned on you signing this authorization. This authorization will expire at the end of the research study unless revoked prior to that time.

VA Boston Healthcare System IRB
Effective Date: April 11, 2022



Version Date: Version 3 (3/16/2022)

| Participant Name: | Date: |
|---|---|
| Title of Study: Highly challenging balance program to reduce fall rate in PD | |
| Principal Investigator: Dr. David Sparrow | VA Facility: VA Boston Healthcare System |

#### WHAT ARE THE COSTS TO ME IF I TAKE PART IN THIS STUDY?

You will not be charged for any treatments or procedures that are part of this study. If you usually pay copayments for VA care and medications, you will still pay these co-payments for VA care and medications that are not part of this study.

Compensation for transportation will be provided by the VA if you require special transportation considerations to travel to the Jamaica Plain campus of the VA Boston Healthcare System. Compensation will be based on total roundtrip mileage at the current GSA mileage rate.

You consent to the release of personally identifying information about you including your name, address, and social security number to the VA so that we may provide compensation to you in the form of a check or debit card. You can expect to receive a check or debit card within 2-6 weeks. The government may garnish the compensation against outstanding debts a veteran has to the federal government.

You consent to the release of personally identifying information about you including your name, address, social security number and bank information (bank name, routing number, and account number) to the VA so that we may provide compensation to you as a direct deposit. You will receive payment within 7 to 10 days.

If payment is made to you by the VA (whether by check, direct deposit, or a VA issued debit card), an IRS Form 1099 will be generated regardless of the amount you are paid.

## WHAT WILL HAPPEN IF I AM INJURED BECAUSE OF MY BEING IN THE STUDY?

If you are injured as a result of taking part in this study, the VA will provide necessary medical treatment at no cost to you unless the injury is due to non-compliance by a study participant with study procedures or if the research is conducted for VA under contract with an individual or non-VA institution.

If you should have a medical concern or get hurt or sick as a result of taking part in this study, call:

DURING THE DAY: Dr. Pantel Vokonas (Medical Director of the VA Normative Aging Study) at 857-364-6400.

AFTER HOURS: Page the person on call for the Normative Aging Study by calling toll free 1-877-204-5849 and ask the answering service to call or page the person on call for the Normative Aging Study

VA Boston Healthcare System IRB
Effective Date: April 11, 2022



Version Date: Version 3 (3/16/2022)

| Participant Name: | Date: |
|---|---|
| Title of Study: Highly challenging balance program to reduce fall rate in PD | |
| Principal Investigator: Dr. David Sparrow | VA Facility: VA Boston Healthcare System |

#### DO I HAVE TO TAKE PART IN THE STUDY?

Your participation in this study is voluntary. If you refuse to take part, you will not suffer any penalty or loss of benefits to which you are otherwise entitled.

You may withdraw from the study at any time. This will end your participation in the study; however, the research team may continue to use the data that have been already collected before your withdrawal. You will be asked to ship all study equipment back to us at no cost to you.

## RIGHT OF INVESTIGATOR TO TERMINATE MY PARTICIPATION

Your participation in the study can be terminated by the study Principal Investigator if it is determined that it is not safe for you to continue in the study. If terminated, you will ship all study equipment back to us at no cost to you.

#### WHO DO I CONTACT ABOUT THIS STUDY IF I HAVE QUESTIONS?

I understand that if I have any medical questions about this research study, I can call Dr. Pantel Vokonas (Medical Director of the VA Normative Aging Study) at (857) 364-6400 during normal working hours.

I understand that if I have any general questions about this research study, I can call Dr. David Sparrow at (857) 364-6400 during normal working hours.

I understand that if I have any medical problems that might be related to this study that during the day I can call Dr. Pantel Vokonas at (857) 364-6400 and after hours I can call toll free 1-877-204-5849 and ask the answering service to call or page the person on call for the Normative Aging Study.

If you have questions about your rights as a study participant or any other questions, complaints, concerns or suggestions about this study, you may contact the Institutional Review Board at (617) 637-3794. This is the Board that oversees all human research at VA Boston Healthcare Systems and has the responsibility to ensure the safety of human participants in this study.

### WILL I BE TOLD NEW INFORMATION ABOUT THIS STUDY?

You will be told of any significant new findings that come to light during the course of this study and that may relate to your wanting to stay in the study.

FOR IRB USE ONLY

VA Boston Healthcare System IRB

Effective Date: April 11, 2022



### AGREEMENT TO PARTICIPATE IN THE RESEARCH STUDY

The study coordinator has explained the research study to you. You have been told of the risks or discomforts and possible benefits of the study. You have been told of other choices of treatment available to you. You have been given the chance to ask questions and obtain answers.

By signing this document below, you voluntarily consent to participate in this study and authorize the use and disclosure of your health information in this study. You also confirm that you have read this consent, or it has been read to you. You will receive a copy of this consent after you sign it.

| I agree to participate in this research study as has been explained in this form. | | |
|---|---|---|
| Participant's Name | Participant's Signature | <br>Date |

FOR IRB USE ONLY